CLINICAL TRIAL: NCT06010849
Title: The Relationship of Trunk Control With Balance, Upper Extremity and Lower Extremity Functions in Stroke Patients
Brief Title: Trunk Control and Extremity Functions in Stroke
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Zekiye İpek KATIRCI KIRMACI, ass. prof, Kahramanmaras Sutcu Imam University
Other Study IDs: ipkkrmc
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: Stroke; Trunk Control; Balance; Function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Trunk control — Trunk control

SUMMARY:
The trunk is the key point of the body. Proximal trunk control is essential for distal extremity movements, balance and functional activities. The aim of the study is to examine the relationship of trunk control with balance, upper extremity and lower extremity functions in stroke patients.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death in developed countries after heart disease and cancer. In adults, it ranks first among neurological diseases in terms of causing death and disability.

About one-third of stroke patients experience permanent physical dysfunction. This situation has a negative impact on the economic, social, psychological life and general quality of life of the patient and his family. Stroke is one of the leading causes of long-term disability in adults due to problems such as activity limitations and participation restrictions caused by disorders in body functions . At this point, rehabilitation in stroke patients has an important place in ensuring the social participation of the patient and minimizing the disorders.

When the literature is examined, it is stated that the best functional results are revealed by a good postural control. Because the trunk is the key point of the body. Proximal trunk control is essential for distal extremity movements, balance and functional activities. It provides trunk control, static and dynamic posture, upright posture of the body, and selective trunk movements .

There are many treatment approaches to increase trunk stabilization. Gaining early trunk control is one of the basic principles of Bobath, which adopts the neurodevelopmental behavior model from neurophysiological approaches.

In recent years, core stabilization exercises, which play an active role in trunk stabilization, have started to be included in the rehabilitation program of stroke patients. Haruyama et al. demonstrated the effectiveness of core stabilization exercises on trunk control, standing, and mobility. This study also indicated the importance of trunk stabilization in balance and mobility (5).

Trunk control means more than just sitting balance. Organization of postural and correction reactions, stability required for the creation of extremity movements, rotation, appropriate gait pattern, proximal stabilization to contribute to distal movement, establishment of the connection between shoulder and pelvis are provided by good trunk control. The trunk, which makes up 60% of our body mass, is necessary for controlling the force created in our body and for optimum movement in the extremities. The holistic system that includes the lower extremities, pelvis, trunk and upper extremities is called the kinetic chain. The creation, collection and transfer of the force required for extremity movements from the lower extremity to the upper extremity are made possible by this system. Thus, these segments, which are independent from each other from proximal to distal, work in a certain interaction and harmony during functional activities (6).

The aim of the study is to examine the effect of trunk control on balance, upper extremity and lower extremity functions in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

-55-85 years old, had an ischemic stroke at least 6 months ago, was at stage 2 according to brunstroma, had a mini-mental test score above 22, could stand independently for 3-4 seconds,

Exclusion Criteraia had orthopedic problems.

Ages: 55 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
The Trunk Impairment Scale | at baseline
  The Trunk Impairment Scale (TIS) consists of 3 parts: 3 items as static sitting balance, 10 items as dynamic sitting balance, and 4 items as coordination. The maximum points received are 7, 10 and 6 points respectively. The total score of TIS is between 0 and 23. High scores indicate good trunk control (6). Turkish validity and reliability study of TIS was also conducted
Berg Balance Scale (BBS) | at baseline
  BBS: It is the gold standard scale that clinically evaluates balance and postural control. It is a 14-item scale that measures the ability to maintain balance while performing functional tasks. Each item is scored between 0 and 4. If the total score is 56 and above, the balance is considered good.
Fugl meyer lower extremity test | at baseline
  FML: It includes subsections that evaluate hip, knee, ankle joint movements, coordination and reflex activities. The highest score that can be obtained from this assessment is 34.
Fugl meyer upper extremity test | at baseline
  FMU: It includes subsections that evaluate joint movements, coordination and reflex activities related to shoulder, elbow, forearm, wrist and hand. The highest score that can be obtained from this assessment is 66.

CONTACTS AND LOCATIONS:
Overall Officials: zekiye ipek katırcı kırmacı, Principal Investigator — kahramanmaras sütçü imam university
Locations (1):
- Kahramanmaraş Sütçü Imam University, Kahramanmaraş, Turkey (Türkiye)